CLINICAL TRIAL: NCT04558749
Title: Assessment of Anxiety and Depression Among Pregnant Women During COVID-19 Pandemic
Brief Title: Anxiety and Depression Among Pregnant Women During COVID-19 Pandemic
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Principal investigator, Assiut University
Other Study IDs: ADCOVID
Record Dates: First submitted 2020-09-18; First posted 2020-09-22 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Psychiatric Status Rating Scales

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: The study population comprised women that will attend their routine visit to the antenatal clinic. The study population will be recruited by using simple random sampling method after verbal consent will be obtained. Resident in the Department of Obstetrics and Gynaecology who will be trained to administer the questionnaire will interview women. Face masks will be provided to the study population during the process of data collection.
  Interventions: Other: State-trait anxiety inventory scale; Other: Edinburgh Postnatal Depression Scale (EDPS)

INTERVENTIONS:
Other: State-trait anxiety inventory scale — This scale is composed of two parts, part one measures anxiety traits and part two measures anxiety state. Each part comprises 20 statements. This scale is a (4) point scale, with a score ranging a minimum of 20 grades to a maximum of 80 grades.
Other: Edinburgh Postnatal Depression Scale (EDPS) — The EPDS is a self-report measure that focuses on the cognitive symptoms of depression. It excludes somatic items that might generate false positives both during pregnancy and after childbirth.7 The EPDS consists of 10 items, each scored 0-3 points, with a potential scale score of 0-30.

SUMMARY:
Pregnancy and early parenthood are life changing periods characterized by intense emotions and a high vulnerability to emotional problems. Overall 10 - 20 % of pregnant women and women in early postpartum period suffer from mental health problems.

In the first months of 2020 , pregnant and breastfeeding women have also needed to face the COVID19 pandemic including the exceptional quarantine measures that have disturbed private and professional life . In addition to the fear of infection , these measures might have negatively impacted the emotional wellbeing of women . As depressive symptoms and anxiety in the pre and peripartum period have been associated with adverse maternal , neonatal and infant outcomes , the psychological impact of COVID19 , and its associated quarantine measures , on pregnant women and new mothers is cause for concern

ELIGIBILITY:
Inclusion Criteria:

All pregnant women presented to the Antenatal care clinic, will be included in the study irrespective of the gestational age of the pregnancy

Exclusion Criteria:

Women previously diagnosed with any psychiatric disorder.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population comprised women that will attend their routine visit to the antenatal clinic. The study population will be recruited by using simple random sampling method after verbal consent will be obtained. Resident in the Department of Obstetrics and Gynaecology who will be trained to administer the questionnaire will interview women. Facemasks will be provided to the study population during the process of data collection.
Sampling Method: Probability Sample
Enrollment: 238 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
The mean scores anxiety and depression among pregnant women during COVID-19 pandemic | one hour
  This scale is composed of two parts, part one measures anxiety traits and part two measures anxiety state. Each part comprises 20 statements. This scale is a (4) point scale, with a score ranging a minimum of 20 grades to a maximum of 80 grades.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No